CLINICAL TRIAL: NCT04519294
Title: A Prospective, Randomized Study to Evaluate the Safety and Effectiveness of Steerable Ureteroscopic Renal Evacuation(SURE)Using the CVAC™ Aspiration System Compared to Basketing for the Removal of Renal Calculi Following Laser Lithotripsy
Brief Title: Comparison of Laser Lithotripsy With and Without Steerable Ureteroscopic Renal Evacuation (SURE)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Calyxo, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP00001
Record Dates: First submitted 2020-08-17; First posted 2020-08-19 (Actual); Results first posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Kidney Stone; Renal Stone; Urolithiasis
MeSH Terms: conditions — Kidney Calculi; Nephrolithiasis; Urolithiasis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- SURE (Active Comparator)
  Interventions: Device: SURE
- Standard Ureteroscopy (Basketing) (Active Comparator)
  Interventions: Device: Standard Ureteroscopy (Basketing)

INTERVENTIONS:
Device: SURE — The SURE stone evacuation procedure is a technique intended to more easily and completely remove a kidney stone during a kidney stone treatment. The urologist first uses a laser to break the kidney stone into small pieces. Then with the SURE procedure, the pieces are gently vacuumed out of the kidney instead of retrieving the pieces one-by-one with a basket or leaving them to pass naturally in the urine. Basketing is allowed and might be used with the SURE procedure, if needed to remove some small stones.
  Arms: SURE
Device: Standard Ureteroscopy (Basketing) — This is a treatment in which the urologist uses a laser to break a kidney stone into small pieces and then uses a tool called a basket to retrieve the pieces one at a time.
  Arms: Standard Ureteroscopy (Basketing)

SUMMARY:
The purpose of the study is to compare the effects, good and/or bad, of a treatment for removing kidney stones called the SURE procedure for stone evacuation to the standard treatment using a basket for stone removal.

ELIGIBILITY:
Inclusion Criteria:

* Candidate for ureteroscopy with laser lithotripsy;
* Presence of renal stone(s);
* Be willing and able to return for all study-related follow up procedures; and,
* Have been informed of the nature of the study, agreeing to its requirements, and have signed the IRB approved informed consent.

Exclusion Criteria:

* BMI > 45;
* Significant comorbidities;
* Bladder, ureteral or kidney abnormalities;
* Pregnant individuals; or
* Unable to meet the treatment and follow up protocol requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2021-06-16 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2025-04-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Mayo Clinic, Phoenix, Arizona
  - Arizona Institute of Urology, Tucson, Arizona
  - Johns Hopkins, Baltimore, Maryland
  - New Jersey Urology, Voorhees Township, New Jersey
  - Albany Medical College, Albany, New York
  - Duke University, Durham, North Carolina
  - Prisma Health, Greenville, South Carolina
  - Urology Austin, Austin, Texas
  - Dell Medical School, The University of Texas at Austin, Austin, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Urology of Virginia, Virginia Beach, Virginia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In total, 132 subject were enrolled and treated. Of the subjects, 123 were randomized. Of these subjects, subjects whose study participation was discontinued prior to the 30-Day CT, who had poor CT quality, major protocol deviations, or who had their procedures aborted were not included in the efficacy analysis. A total of 101 subjects qualified for the efficacy analysis.
Period: Overall Study
Arm/Group | SURE | Standard Ureteroscopy (Basketing)
Started | 46 | 55
Completed | 43 | 50
Not Completed | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SURE | Standard Ureteroscopy (Basketing) | Total
Number analyzed (Participants) | 46 | 55 | 101
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 59 (14) | 60 (14) | 59 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 27 | 49
  Male | 24 | 28 | 52
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White (Not Hispanic) | 36 | 44 | 80
  Black or African American | 2 | 5 | 7
  Hispanic/Latino | 7 | 6 | 13
  Asian | 1 | 0 | 1
Total stone burden [Mean (Standard Deviation); unit: mm] | 14 (6.5) | 19 (11) | 17 (9)
Total stone volume [Mean (Standard Deviation); unit: mm^3] | 490 (430) | 710 (560) | 610 (510)

OUTCOME MEASURES:

1. Primary Outcome: Stone Free Rate (SFR) - Zero Fragments
Description: The primary efficacy endpoint is the SFR, where stone free status is defined as zero residual fragments at 30 days observed on non-contrast CT (NCCT) (1.25mm slice thickness) by blinded central reviewer(s). The SFR is calculated by determining the number of subjects in each treatment arm with a stone free status of zero fragments and dividing that by the total number of subjects treated in the respective treatment arm.
Time Frame: 30 Days
Population: All patients who met all protocol requirements with no major deviations that compromise the ability to assess primary and secondary endpoints.
Measure: Number; unit: % subjects
Groups:
- Standard Ureteroscopy (Basketing): This is a treatment in which the urologist uses a laser to break a kidney stone into small pieces and then uses a tool called a basket to retrieve the pieces one at a time.
  Other Name:
Arm/Group | SURE | Standard Ureteroscopy (Basketing)
Number analyzed (Participants) | 46 | 55
% subjects | 48 | 49

2. Secondary Outcome: Residual Stone Volume (RSV)
Description: A continuous quantitative measure of remaining stone volume following intervention, assessed via post-procedural imaging on NCCT (1.25mm slice thickness) by blinded central reviewer(s).
Time Frame: 30 Days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | SURE | Standard Ureteroscopy (Basketing)
Number analyzed (Participants) | 46 | 55
mm^3 | 14.3 (30.9) | 70.2 (144.9)

3. Secondary Outcome: Stone Clearance (% Reduction in Stone Volume)
Description: Percent reduction ([Baseline stone volume- 30-Day stone volume] / Baseline stone volume) in stone volume following intervention, assessed via post-procedural imaging on NCCT (1.25mm slice thickness) by blinded central reviewer(s).
  A positive result indicates a decrease in stone volume removed during the procedure; a negative value indicates an increase in stone volume following the procedure.
Time Frame: 30 Days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent reduction (%)
Arm/Group | SURE | Standard Ureteroscopy (Basketing)
Number analyzed (Participants) | 46 | 55
percent reduction (%) | 97.1 (5.4) | 93.3 (11.7)

ADVERSE EVENTS:
Time Frame: 30 Day
Description: Reporting adverse events per requirements per the Results Data Element Definitions.
Arm/Group | SURE | Standard Ureteroscopy (Basketing)
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/65
Serious Adverse Events (participants affected / at risk) | 1/67 | 2/65
Other Adverse Events (participants affected / at risk) | 4/67 | 5/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SURE (N=67) | Standard Ureteroscopy (Basketing) (N=65)
Sepsis Requiring Hospitalization (Renal and urinary disorders) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SURE (N=67) | Standard Ureteroscopy (Basketing) (N=65)
Ureteral Damage (Renal and urinary disorders) | 4 (4) | 5 (5) — Clavien-Dindo Grade I

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-26): https://cdn.clinicaltrials.gov/large-docs/94/NCT04519294/Prot_SAP_000.pdf